CLINICAL TRIAL: NCT03798574
Title: The Long-term Impact of Invasive Meningococcal Disease in Australian Adolescents and Young Adults
Acronym: AMEND
Status: Completed | Type: Observational
Sponsor: University of Adelaide (Other)
Responsible Party: Principal Investigator, Helen Marshall, Professor, University of Adelaide
Other Study IDs: HREC/14/WCHN/024
Record Dates: First submitted 2018-12-23; First posted 2019-01-10 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Meningococcal Infections; Neisseria Meningitis Sepsis; Neisseria Infection
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IMD Case: No intervention
- Control: No intervention

SUMMARY:
Survivors of invasive meningococcal disease (IMD) experience a range of mild to severe sequelae that impact upon their quality of life. The majority of studies to date have focused on the impact of IMD on childhood and very little is known about the impact of the disease on adolescents and young people.

The aim of this study is to assess the physical, neurocognitive, economic and societal impact of IMD on adolescents and young adult Australian survivors.

Hypothesis:

1. Adolescents and young adult survivors who are 2 to 10 years post IMD have significantly poorer outcomes including intellectual functioning and quality of life when compared to healthy controls.
2. IMD imposes a significant financial burden upon individuals, families and society.
3. Serogroup B disease is associated with an increased risk of sequelae when compared to non-B serogroup IMD.

Study design:

This a multi-centre, case-control mixed-methods study. Survivors of IMD (retrospective and prospective cases) and non-IMD healthy controls will be invited to participate in the study.

Retrospective IMD cases admitted in the previous 10 years will be identified through each of the participating hospitals (paediatric and adult hospitals). During the course of the study prospective recruitment of IMD cases will also occur at participating hospitals. Meningococcal foundations/groups will also be approached and asked to advertise and conduct a mail out to their members to inform them about the study.

Healthy controls will be prospectively recruited by "snowballing technique" whereby enrolled IMD cases will be asked to distribute a study information sheet to their healthy friends/acquaintances who are approximately the same age. Control participants may also be identified from databases at each participating site or through community advertising.

Enrolled cases will undergo a neurocognitive, psychological and physical examination 2 - 10 years post IMD admission. A subset of IMD cases will be invited to participate in a semi-structured interview. Controls will also undergo neurocognitive, psychological and physical examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 15 to 24 years 11 months at time of IMD admission
* Hospitalised IMD case from 1st January 2006 -with serogroup B or non-B IMD, confirmed by culture or polymerase chain reaction (PCR) in blood or CSF.
* Healthy controls aged 17 to 34 years 11 months at the time of assessment.

Exclusion Criteria:

* Individuals who are not fluent with the English language.
* Control participants with a history of meningitis, encephalitis, or meningococcal disease, intellectual disability, intracranial pathology (eg. traumatic brain injury) that may impact on cognitive functioning, or significant vision and/or hearing loss that may impact on the validity or reliability of the neurocognitive assessment.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Population sample from participating Australian hospitals in Adelaide, Melbourne, Perth, and Sydney.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Difference in intellectual functioning between cases and controls | Between 2 to 10 years post IMD admission
  Measured by the Full Scale intelligence quotient (IQ) score obtained from the Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV)
Difference in quality of life between cases and controls | Between 2 to 10 years post IMD admission
  Measured by the overall multi-attribute health utility score obtained from the Health Utilities Index Mark 3 (HUI3)-15Q self-report.

SECONDARY OUTCOMES:
Difference in academic achievement between cases and controls. | Between 2 to 10 years post IMD admission
  Measured by Wechsler Individual Achievement Test - Second Edition (WIAT-II)
Difference in memory (verbal and visual) between cases and controls. | Between 2 to 10 years post IMD admission
  Measured by Verbal Learning and Design Memory subtests from the Wide Range Assessment of Memory and Learning, Second Edition (WRAML2)
Difference in executive functioning between cases and controls. | Between 2 to 10 years post IMD admission
  Measured by Delis-Kaplan Executive Function System (D-KEFS)
Difference in executive functioning between cases and controls assessed through BRIEF self-report questionnaire | Between 2 to 10 years post IMD admission
  Assessed through BRIEF self-report questionnaire (parent and/or self-report)
Difference in the frequency of psychiatric disorders between cases and controls. | Between 2 to 10 years post IMD admission
  Assessed through Mini International Neuropsychiatric Interview (M.I.N.I 6.0)
Difference in psychological functioning between cases and controls. | Between 2 to 10 years post IMD admission
  Assessed through self report questionnaire Depression Anxiety Stress Scales (DASS) (self-report)
Difference in behavioral ratings between cases and controls | Between 2 to 10 years post IMD admission
  Measured by Conners Rating Scales (parent and/or self-report)
Difference in health and disability functioning between cases and controls | Between 2 to 10 years post IMD admission
  Measured by the International Classification of Functioning, Disability and Health (ICF) tool.
Difference in hearing threshold levels between cases and controls | Between 2 to 10 years post IMD admission
  Measured by pure tone audiometry.
Difference in health status between cases and controls | Between 2 to 10 years post IMD admission
  The EQ-5D-5L will be completed to measure participant's health status and to calculate quality adjusted life years (QALYS) lost.
To estimate the lifetime costs associated with survival following IMD | From time of admission up to time of follow up (2 to 10 years post IMD admission)
  IMD cases only: Lifetime dollar costs.
Explore adolescents and young people's experience of their hospital presentation, admission, and recovery from IMD | Between 2 to 10 years post IMD admission
  A subset of IMD cases will participate in a semi-structured interview.
Carer's experience assessed through the Carer Experience Scale | Between 2 to 10 years post IMD admission
  For those IMD cases with a disability, the primary caregiver and other family members living in the same household will be invited to complete the Carer Experience Scale.
Carer's experience assessed through ICEpop CAPability questionnaires | Between 2 to 10 years post IMD admission
  For those IMD cases with a disability, the primary caregiver and other family members living in the same household will be invited to complete ICEpop CAPability questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Marshall, Principal Investigator — University of Adelaide
Locations (4):
- Australia (4):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Women's and Children's Hosptial, Adelaide, South Australia
  - Monash Children's Hospital, Melbourne, Clayton, Victoria
  - Perth Children's Hospital, Nedlands, Western Australia

REFERENCES:
- [Derived] Marshall H, McMillan M, Wang B, Booy R, Afzali H, Buttery J, Blyth CC, Richmond P, Shaw D, Gordon D, Barton B. AMEND study protocol: a case-control study to assess the long-term impact of invasive meningococcal disease in Australian adolescents and young adults. BMJ Open. 2019 Dec 29;9(12):e032583. doi: 10.1136/bmjopen-2019-032583. PMID 31888931